CLINICAL TRIAL: NCT05496829
Title: IMPACT Trial: Intervention to iMProve AdherenCe Equitably
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Dawn L. Hershman, Assistant Professor of Medicine, Division of Hematology/Oncology, Columbia University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAT8817; 1P50MD017341 (NIH)
Record Dates: First submitted 2022-06-17; First posted 2022-08-11 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adherence Intervention (Experimental): Multicomponent Adherence Intervention
  Interventions: Behavioral: Multicomponent Adherence Intervention
- Usual Care (Other): Usual Care from treating providers
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Multicomponent Adherence Intervention — The adherence intervention will be comprised of a participant preference approach in which all participants undergo a baseline pharmacist-led medication optimization session and are offered training in how to use the patient portal and freely-available smartphone reminder app.
  Arms: Adherence Intervention
Other: Usual Care — Receipt of usual care from providers
  Arms: Usual Care

SUMMARY:
To determine the efficacy of a multicomponent adherence intervention among participants with early-stage breast cancer on endocrine therapy and at least one oral cardiovascular disease (CVD) medication on adherence to endocrine therapy and to CVD medication at 24 weeks assessed by self-report using the Domains of Subjective Extent (DOSE)-Nonadherence questionnaire and also by pharmacy fill data assessed in the electronic health record (EHR).

ELIGIBILITY:
Inclusion Criteria:

* Women or men age >18 years
* Diagnosed with stage I-III breast cancer prescribed endocrine therapy
* Within 3-years of the end of early active treatment (e.g., surgery, chemotherapy not including human epidermal growth factor receptor 2 (HER2)-directed therapy, radiation)
* Patients must be prescribed at least 1 antihypertensive or statin medication for CVD prevention
* Self-report of at least some nonadherence ET or CVD medication on DOSE-Nonadherence Extent of Nonadherence questionnaire

Exclusion Criteria:

* Evidence of breast cancer recurrence
* Non-English or Non-Spanish speaking
* Not cognitively able to complete study requirements
* Do not follow with either a primary care provider or cardiologist within the New York Presbyterian Health system's Epic EHR
* Inability to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Adherent to Endocrine Therapy (ET) and CVD Medication at 24 Weeks | 24 Weeks
  Adherence to ET and CVD medication is a composite of both medication refills at 24 weeks (proportion of days covered (PDC) ≥80%) and self-report of taking the medication (as per DOSE-Nonadherence questionnaire; 3-item questionnaire in which participants with perfect adherence on each item will be categorized as adherent). Participants will be categorized as adherent if they have medication available by pharmacy fills and report being adherent to taking their pills day-today via self report.

SECONDARY OUTCOMES:
Number of Participants Adherent to ET and CVD Medication at 52 Weeks | 52 Weeks
  Adherence to ET and CVD medication is a composite of both medication refills at 52 weeks (proportion of days covered (PDC) ≥80%) and self-report of taking the medication (as per DOSE-Nonadherence questionnaire; 3-item questionnaire in which participants with perfect adherence on each item will be categorized as adherent). Participants will be categorized as adherent if they have medication available by pharmacy fills and report being adherent to taking their pills day-today via self report.
Change in blood pressure at 24 weeks | Baseline to 24 weeks
  To compare office blood pressure changes from baseline to 24 weeks
Change in blood pressure at 52 weeks | Baseline to 52 weeks
  To compare office blood pressure changes from baseline to 52 weeks
Change in low-density lipoprotein (LDL) cholesterol | Baseline to 52 weeks
  To compare changes in low-density lipoprotein (LDL) cholesterol from baseline to 52 weeks.
Changes in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 at 24 weeks | Baseline and 24 weeks
  To evaluate changes in healthcare related quality of life (HRQOL), measured by the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 at baseline and 24 weeks. The Patient-Reported Outcomes Measurement Information System (PROMIS) 29 is a well-validated assessment tool that includes 29 questions evaluating 7 domains including physical function, anxiety, depression, fatigue, sleep, social functioning, and pain interference (which is often associated with ET adherence). Several of these measures have been important determinants of medication adherence and have the potential to moderate intervention effects.
Changes in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 at 52 weeks | Baseline and 52 weeks
  To evaluate changes in healthcare related quality of life (HRQOL), measured by the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 at baseline and 52 weeks. The Patient-Reported Outcomes Measurement Information System (PROMIS) 29 is a well-validated assessment tool that includes 29 questions evaluating 7 domains including physical function, anxiety, depression, fatigue, sleep, social functioning, and pain interference (which is often associated with ET adherence). Several of these measures have been important determinants of medication adherence and have the potential to moderate intervention effects.
Changes in Treatment Satisfaction Questionnaire for Medication (TSQM) at 24 Weeks | Baseline and 24 weeks
  To compare participants' satisfaction with their medication regimens as measured by the Treatment Satisfaction Questionnaire for Medication (TSQM). The 14-item TSQM Version 1.4 is a reliable and valid instrument to assess participants' satisfaction with medication, providing scores on four scales - side effects, effectiveness, convenience and global satisfaction.
Changes in Treatment Satisfaction Questionnaire for Medication (TSQM) at 52 Weeks | Baseline and 52 weeks
  To compare participants' satisfaction with their medication regimens, as measured by the Treatment Satisfaction Questionnaire for Medication (TSQM). The 14-item TSQM Version 1.4 is a reliable and valid instrument to assess participants' satisfaction with medication, providing scores on four scales - side effects, effectiveness, convenience and global satisfaction.
Changes in Medical Adherence Self-Efficacy Scale (MASES) at 24 Weeks | Baseline and 24 weeks
  To compare participants' self-efficacy with their medication regimens as measured by the Medical Adherence Self-Efficacy Scale (MASES) at baseline and 24 weeks. MASES is a 13-item form, 12 of the items ask about confidence in ability to make medication adherence part of daily routine. The total scale ranges from 1-4, and it is an average score of all 13 items.
Changes in the Medical Adherence Self-Efficacy Scale (MASES) at 52 Weeks | Baseline and 52 weeks
  To compare participants' self-efficacy with their medication regimens as measured by the Medical Adherence Self-Efficacy Scale (MASES) at baseline and 52 weeks. MASES is a 13-item form, 12 of the items ask about confidence in ability to make medication adherence part of daily routine. The total scale ranges from 1-4, and it is an average score of all 13 items.
Change in Regimen Complexity | Baseline and at 52 weeks
  To evaluate regimen complexity at baseline and at 52 weeks. This will be extracted through manual chart review from the EHR. The investigators will extract total number of prescription medications and frequency of dosing for CVD medications as ET is once daily.
Subject reasons using the DOSE-Nonadherence reasons for nonadherence questionnaire | at baseline
  To evaluate reasons for medication nonadherence at baseline using the DOSE-Nonadherence reasons for nonadherence questionnaire
Reasons for Medication Non-adherence using the DOSE-Nonadherence Reasons for Nonadherence Questionnaire at 24 Weeks | 24 weeks
  To evaluate reasons for medication nonadherence at 24 weeks using the DOSE-Nonadherence reasons for nonadherence questionnaire. The DOSE-Nonadherence Reasons for Nonadherence questionnaire asks how much 21 reasons for nonadherence contribute to missing doses such as trouble affording medications, insufficient social support, complexity of regimen, and concerns about adverse effects. This will be used to assess the effect of the intervention on barriers to adherence.
Reasons for Medication Non-adherence using the DOSE-Nonadherence Reasons for Nonadherence Questionnaire at 52 Weeks | 52 weeks
  To evaluate reasons for medication nonadherence at 52 weeks using the DOSE-Nonadherence reasons for nonadherence questionnaire. The DOSE-Nonadherence Reasons for Nonadherence questionnaire asks how much 21 reasons for nonadherence contribute to missing doses such as trouble affording medications, insufficient social support, complexity of regimen, and concerns about adverse effects. This will be used to assess the effect of the intervention on barriers to adherence.
Impact of events using the Impact of Events Scale (IES) | Baseline
  To evaluate the impact of events using the Impact of Events Scale (IES) to evaluate intrusive and avoidant thoughts about participant's underlying breast cancer diagnosis at baseline. IES is a 15-item scale which queries intrusive and avoidant thoughts about a distressing event (breast cancer) in the past 7 days (similar to post-traumatic stress disorder [PTSD] symptoms). Each item has a scoring range of 0 (not at all)-5(often). This scale has been associated with disparities in ET and CVD medication nonadherence

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sathe C, DeStephano D, Lee S, West H, Beauchemin M, Accordino M, Liyanage-Don N, Crew KD, Kukafka R, Harden E, Hershman DL, Kronish IM. Rationale and design of the IMProving Adherence to medications for breast Cancer and cardiovascular disease equiTably (IMPACT) randomized clinical trial. Contemp Clin Trials. 2025 Sep;156:108009. doi: 10.1016/j.cct.2025.108009. Epub 2025 Jul 11. PMID 40653311